CLINICAL TRIAL: NCT06854016
Title: Randomized, Sham Controlled, Single Blind Study on the Performance and Safety of Photo Biomodulation Therapy (PBMT) With LightForce® Therapy Lasers on Lateral Ankle Sprain Pain Reduction
Brief Title: Performance and Safety of LightForce® Therapy Lasers on Lateral Ankle Sprain
Acronym: BRIGHT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DJO UK Ltd (Industry)
Collaborators: Donawa Lifescience Consulting SRL (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENOVIS-S-INP-0011
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Ankle Sprain 1St Degree; Ankle Sprain 2Nd Degree; Acute Pain
Keywords: lateral acute grade I and II ankle sprain, pain, laser
MeSH Terms: conditions — Acute Pain; Pain | interventions — Laser Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Laser treatment - Arm 1 (Sham Comparator): Sham Laser therapy
  Interventions: Device: Sham Laser therapy; Other: RICE and physiotherapy/exercise protocol
- Laser Treatment - Arm 2 (Active Comparator): Laser therapy
  Interventions: Device: Laser therapy; Other: RICE and physiotherapy/exercise protocol

INTERVENTIONS:
Device: Sham Laser therapy — sham laser therapy for 4 consecutive weeks with a minimum of 3 sessions per week, for the first 2 weeks, and then a minimum of 2 sessions per week for the following 2 weeks.
  Arms: Sham Laser treatment - Arm 1
Device: Laser therapy — laser therapy for 4 consecutive weeks with a minimum of 3 sessions per week, for the first 2 weeks, and then a minimum of 2 sessions per week for the following 2 weeks.
  Arms: Laser Treatment - Arm 2
Other: RICE and physiotherapy/exercise protocol — RICE plus physiotherapy/exercise protocol represents the standard of care (SOC) and the program includes: for the first 2 weeks RICE protocol performed daily at home by the patient, for the following 4 weeks a physiotherapy/exercise protocol will be performed at site with 2 sessions per week.

SUMMARY:
DJO UK Ltd (ENOVIS) is conducting this study to assess the effectiveness of LightForce® Therapy Lasers on pain reduction in subjects with ankle soft tissue trauma and/or sport injury. In detail this study will assess superiority of LightForce® Therapy Lasers combined with standard of care, represented by RICE and physiotherapy/exercise program, compared to sham laser combined with standard of care (RICE and physiotherapy/exercise program) on pain reduction in subjects with acute grade I - II lateral ankle sprain. In addition, this study allows to collect post market clinical data on the safety and performance of LightForce® Therapy Lasers, when used, following the normal clinical practice, in accordance with its approved and CE marked intended use.

DETAILED DESCRIPTION:
This clinical investigation is a post-market, International, multi center, prospective, randomized, sham controlled, single blind study to assess the effectiveness of LightForce® Therapy Lasers and to collect PMCF data on the safety and performance of LightForce® Therapy Lasers when used in accordance with its approved labeling, to comply with Medical Device Regulation (EU) 2017/745 (MDR) Article 61 and Part B of Annex XI.

ELIGIBILITY:
Inclusion Criteria:

1. Patient male or female with age ≥18 years old
2. Patient with diagnosis of LAS (as confirmed by physical examination) to be treated by LightForce® Therapy Lasers according to its indications.
3. Patient suffering from LAS pain for no more than 72 hours prior to enrollment
4. Pain (either persistent or during activities) score reported by the subject at baseline ≥ 40 mm measured on VAS
5. Patient able to provide written informed consent

Exclusion Criteria:

1. Patient with musculoskeletal pathological conditions not to be treated with/contraindication to the use of LightForce® Therapy Lasers according to its intended use and indications
2. Patients who are taking drugs that have heat or light sensitive contraindications, such as but not limited to certain types of steroids
3. Patients who have been administered with corticosteroids after injury
4. Pregnant females or females of childbearing potentially planning to become pregnant during the study participation
5. Patients who had systemic inflammatory conditions (i.e. rheumatoid arthritis, polymyalgia rheumatica)
6. Patients affected by chronic ankle instability (recurrent sprains, ankle instability, functional ankle instability, mechanical ankle instability fol¬lowing the first-time injury)
7. Patients with bilateral ankle sprain
8. Patients who have a disease that would limit their participation in exercises (i.e. severe chronic obstructive pulmonary disease, severe heart failure, cerebrovascular event history)
9. Patients with fractures (as confirmed by radiological examination)
10. Patients with a diagnosis of active cancer
11. Patients with tattoos covering more than 30% of the area to be treated with LightForce® Therapy Lasers
12. Patients who are mentally or physically incapacitated
13. Patient participating in other clinical study or has completed a clinical study less than 30 days prior to enrollment
14. Patients with other clinically significant co-morbidities that make the patient unsuitable for study participation, at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Pain change | 2 weeks after treatment start
  Pain reduction measured with Visual Analog Scale (VAS) (in a scale 0-100 mm, where 0 is no pain and 100 is the worst possible pain) after 4 weeks of treatment compared to pre-treatment (baseline) VAS

SECONDARY OUTCOMES:
Safety - adverse event rate | through study completion, an average of 12 weeks
  Proportion of patient experiencing an adverse event associated with device use

OTHER OUTCOMES:
Pain change | 1,3,4, 6 and 12 weeks after treatment start
  Pain measured with Visual Analog Scale (VAS) (in a scale 0-100 mm, where 0 is no pain and 100 is the worst possible pain) at 1,3,4, 6 and 12 weeks after treatment start to assess short-term and long-term pain management compared to baseline
Ankle pain and Disability | 1, 2, 3, 4, 6 and at 12 weeks after treatment start
  Ankle pain and disability measured with the Foot and Ankle Disability Index (FADI) questionnaire (the score output is given as a percentace) and the highest the percentage the better is the clinical outome, the lowest the percentage the worse is the clinical outcome; performed at 1, 2, 3, 4, 6 and at 12 weeks after treatment start compared to baseline.
Patient overall status change | 2, 4, 6 ans 12 weeks after treatment start
  Patient ratings of overall improvement, assessed by QoL (SF-12): The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. The SF-12 uses 12 items and scores range from 0 to 100, with higher scores indicating better physical and mental health functioning. SF-12 will be assessed at 2, 4, 6 weeks and at 12 weeks and compared to baseline
Range of motion (ROM) of the ankle | 1, 2, 3, 4, 6 and 12 weeks after treatment start
  Range of motion for the ankle (flex-extension) measured by a universal goniometer at 1,2, 4, 6 and 12 weeks after treatment start compared to baseline
Return to pre-injury activity/sport level | 2, 3, 4, 6 and 12 weeks after treatment start
  Return to pre-injury activity/sport level measured on a 1 to 5 Likert scale at 2, 3, 4 ,6 and 12 weeks. This will be assessed as time-to-recovery: time after injury needed for the patient to reach the pre injury/sport level.

CONTACTS AND LOCATIONS:
Overall Officials: Ove Indergaard, Physiotherap, Principal Investigator — ove@indergaardphysio.com
Locations (8):
- Italy (6):
  - Carioni Fisioterapia, Cassano d'Adda, Milano
  - Casertafisio, Caserta
  - Rachis Center, Roma
  - Fisiolab3, Roma
  - Fisioterapia Eur, Roma
  - Fisioterapia Gardenie, Roma
- United Kingdom (2):
  - INDERGAARD PHYSIOTERAPY Ltd, Leeds
  - Freedom Care Clinics, Manchester